CLINICAL TRIAL: NCT04415606
Title: A Pre-Market, Prospective, Controlled, Multicenter, Single Blinded, Pivotal Clinical Investigation of QuikClot Control+ for Use in Mild to Moderate Bleeding
Brief Title: QuikClot Control+ Hemostatic Dressing Use in Mild to Moderate Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Z-Medica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZM-QCC-01
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Hemostasis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subject will not know which arm they were randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- QuikClot Control+ (Experimental): QuikClot Control+
  Interventions: Device: QuikClot Control+
- Standard gauze (Placebo Comparator): Standard gauze per standard of care
  Interventions: Device: QuikClot Control+

INTERVENTIONS:
Device: QuikClot Control+ — Non-absorbable, sterile, X-ray detectable non-woven dressing impregnated with kaolin.

SUMMARY:
QuikClot Control+ Hemostatic Dressing (QuikClot+) is indicated for temporary control of internal organ space bleeding for patients displaying Class III or Class IV Bleeding. It may also be used for control of severely bleeding wounds such as surgical wounds and traumatic injuries. QuikClot Control+ is also indicated for temporary control of mild to moderate bleeding in cardiac surgical procedures. QuikClot Control+ is also indicated for use to control bleeding from bone surface following sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* Age range greater than or equal to 18 years old
* Willing and able to give prior written informed consent
* Requiring cardiac surgery

Exclusion Criteria:

* Subject undergoing emergency surgery for any reason
* Subject has active or potential infection at the surgical site or endocarditis
* eGFR less that lo mL per minute
* Subject who is currently participating in an investigational drug or another device trial (excluding registries)
* Leucopenia (WBC < 3.5x 103/µL), or acute anemia (Hgb < 10.0 mg/dL or 6 mmol/L), or thrombocytopenia (platelet count < 50x 103/µL), or history of bleeding diathesis or coagulopathy, or HIT positive
* Other medical, social, or psychological conditions that, in the opinion of the Investigator, precludes the subject from appropriate consent or adherence to the protocol required follow-up exams
* Active illicit drug use, verbally confirmed with the patient
* Severe Liver dysfunction confirmed via Child-Pugh of B-C or MELD > 10
* Female who is pregnant at screening. Confirmation by urine or serum pregnancy test
* Incarcerated or unable to give voluntary informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Achievement of hemostasis | Up to 10 minutes
  The primary effectiveness endpoint is the rate at which subjects achieve hemostasis (grade 0 bleed) through up to 10 minutes of application and compression of the bleeding site.

SECONDARY OUTCOMES:
Achievement of hemostasis | Up to 5 minute and 10 minutes
  Proportion of subjects achieving hemostasis (grade 0 bleed) measured at 5 minute and 10 minutes of application and compression at the bleeding site.

CONTACTS AND LOCATIONS:
Overall Officials: Mumashir Mumtaz, MD, Principal Investigator — UPMC Pinnacle
Locations (7):
- United States (7):
  - University of Colorado Health, Aurora, Colorado
  - Emory, Atlanta, Georgia
  - Portneuf Medical Center / Snake River Research PLCC, Pocatello, Idaho
  - Washington University, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - UPMC Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided